CLINICAL TRIAL: NCT03872908
Title: Prospective Monocentric Study Evaluating Patients' Satisfaction and Efficacy of Compression Using Surgical Gloves in Peripheral Neuropathies Induced by Taxane or Platinum-based Chemotherapies
Brief Title: Satisfaction & Efficacy of Compression Using Surgical Gloves in Chemo-induced Peripheral Neuropathies
Acronym: ELEGANT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Other Study IDs: ELEGANT - ET18-262
Record Dates: First submitted 2019-03-08; First posted 2019-03-13 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer; Colorectal Cancer
Keywords: Breast cancer; Colorectal cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms | interventions — Gloves, Surgical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Evaluation of patient's satisfaction when wearing surgical gloves (dominant hand) versus chilled gloves (non-dominant hand) at the end of paclitaxel administration.
  Interventions: Device: Chilled gloves; Device: Surgical gloves
- Cohort 2: Evaluation of the efficacy of the compression induced by surgical gloves against peripheral neuropathies in patients treated by oxaliplatine after a 595 mg/m2 cumulated dose.
  Interventions: Device: Surgical gloves

INTERVENTIONS:
Device: Chilled gloves — Chilled glove for non-dominant hand (patients treated with paclitaxel)
  Groups: Cohort 1
Device: Surgical gloves — Surgical gloves (patients treated with oxaliplatine)

SUMMARY:
Evaluation of Satisfaction & Efficacy of Compression Using Surgical Gloves in Peripheral Neuropathies Due to Chemotherapy

DETAILED DESCRIPTION:
Peripheral neuropathy (PN) is an adverse event of numerous chemotherapy agents commonly used, including taxanes (paclitaxel, docetaxel) and platinum-based treatments (oxaliplatine, cisplatine, carboplatine).

Taxanes are widely used in breast cancer. Docetaxel and paclitaxel became indispensable during the last decade in metastatic and early stage breast cancer treatment. For platinum-based chemotherapies, oxaliplatine is one of the main molecules used in digestive oncology, particularly in colorectal cancer.

The limiting toxicities of taxanes and platinum-based treatments which can lead to the therapeutic scheme modification (therefore to a potential diminution of efficacy and eventually to treatment stop) are mainly hematologic (neutropenia) and neurological, the most frequent neuro-toxicity event being a PN associated or not to neuropathic pains. The PN induced by chemotherapy can occur prematurely during the treatment course, persist between the treatments' cycles and last a long time after the end of cycles, with an impact on patients' quality of life. Symptoms are mainly sensitive, including pain, paresthesia and hands / foot numbness. These symptoms, as the hematologic toxicity, represent a major limiting factor for the treatment.

According to the ASCO recommendations, there is no effective prophylactic method against the chemo-induced PN. In a retrospective study, the chilled gloves used for preventing the nail lesions during chemotherapy may reduce the incidence of docetaxel-induced PN. Recently, the surgical gloves efficacy against paclitaxel-induced PN has been evaluated prospectively in women presenting a metastatic or early stage breast cancer, with a percentage of grade >=2 NP significantly lower for the hand protected by surgical gloves than the control hand without glove (compression-induced vasoconstriction responsible for a blood flow reduction in the hands and therefore for the local exposure to chemotherapy agents) and a good tolerance.

Chilled gloves, which use the same principle of vasoconstriction through cold, are also used in the current practice for preventing the PN occurrence. However, contrary to surgical gloves, they can be not well tolerated since the very first cycles (intolerance to cold sensation).

The objective of this study is to evaluate the medium and long term efficacy of compression induced by surgical gloves against the PN development in two frequent indications in oncology, patients treated with paclitaxel (breast cancer) or oxaliplatine (colorectal cancer) and patients' satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years old
* Breast cancer requiring a treatment by paclitaxel or colorectal cancer requiring a treatment by oxaliplatine
* At least 8 chemotherapy cycles planned
* Able to understand, read and write French language
* Covered by a social insurance
* Dated and signed informed consent

Exclusion Criteria:

* Pre-existing neuropathy or history of neuropathy
* Psychological, family, sociological or georgraphical condition that may potentially compromise the adherence to study protocol and follow up
* Cohort 1: Patients presenting a Raynaud's syndrome (contra-indication to cold temperatures)
* Participation to clinical trial which may interfere with the evaluation of the main endpoints.
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with adjuvant or metastatic:
  * Breast cancer treated by Paclitaxel or,
  * Colorectal cancer treated by Oxaliplatine
Sampling Method: Non-Probability Sample
Enrollment: 177 (Actual)
Dates: Start 2019-09-29 (Actual); Primary Completion 2024-02-29 (Estimated); Study Completion 2024-02-29 (Estimated)

PRIMARY OUTCOMES:
Cohort1:Evaluation of patient's satisfaction when wearing surgical gloves (dominant hand) and chilled gloves (non-dominant hand) at the end of paclitaxel administration. | At the end of paclitaxel administration (4 to 6 months after inclusion)
  Global patient's satisfaction evaluated for each hand using a numeric scale from 0 (very unsatisfied) to 10 (very satisfied)
Cohort 2: Efficacy of compression induced by surgical gloves vs peripheral neuropathies development in patients treated by oxaliplatine after a cumulative dose of 595 mg/m2 | After the end oxaliplatine administration (4 to 6 months after inclusion)
  Percentage of NP grade >= 2 after a cumulative dose of 595 mg/m2 using NCI-CTCAE v5

SECONDARY OUTCOMES:
Cohort 1: Evaluation of comfort and pain felt with gloves for each hand | At the end of each cycle (each cycle is 7 days)
  Evaluation using a numeric scale from 0 (Very uncomfortable / Painful) to 10 (Very comfortable / No pain)
Evaluation of the ease to put on gloves for each hand | At the end of paclitaxel administration (4 to 6 months)
  Evaluation using a numeric scale from 0 (Very difficult / long) to 10 (Very easy / Fast)
Cohort 1: Evaluation of the percentage of motor and sensitive peripheral neuropathies for each hand | Before each cycle (except the 1st one), (each cycle is 7 days)
  Evaluation using NPSI and MRC questionnaires
Cohort 1: Evaluation of the percentage of motor and sensitive peripheral neuropathies for each hand | At the end of paclitaxel administration (4 to 6 months after inclusion)
  Evaluation using NPSI and MRC questionnaires
Cohort 1: Evaluation of the percentage of motor and sensitive peripheral neuropathies for each hand | 12 months after the end of treatment
  Evaluation using NPSI and MRC questionnaires
Cohort 1: Evaluation of the percentage of peripheral neuropathies >= 2 for each hand | Before each cycle (except the 1st one) (each cycle is 7 days)
  Evaluation using the NCI-CTCAE v5 scale
Cohort 1: Evaluation of the percentage of peripheral neuropathies >= 2 for each hand | At the end of paclitaxel administration (4 to 6 months after inclusion)
  Evaluation using the NCI-CTCAE v5 scale
Cohort 1: Evaluation of the percentabe of onycholysis grade 2 for each hand | At the end of paclitaxel administration (4 to 6 months after inclusion)
  Evalutation using NCI-CTCAE v5 scale
Cohort 1: Evaluation of nurses's preference for the gloves wearing (surgical versus chilled gloves) | At the end of paclitaxel administration (4 to 6 months after inclusion)
  Evaluation using a numeric scale from 0 (Very xxxx) to 10 (Very xxxx)
Cohort 2: Evaluation of the global satisfaction concerning surgical gloves wearing, comfort, pain and ease to wear | At the end of oxaliplatine administration (4 to 6 months after inclusion)
  Evaluation using a numeric scale from 0 (Very unsatisfied) to 10 (Very satisfied)
Cohort 2: Evaluation of the acute sensitive peripheral neuropathies for each hand | Before each cycle (except the 1st one) (each cycle is 7 days)
  Evaluation using a duration questionnaire
Cohort 2: Evaluation of the acute sensitive peripheral neuropathies for each hand | At the end of oxaliplatine administration (4 to 6 months after inclusion)
  Evaluation using a duration questionnaire
Cohort 2: Evaluation of the peripheral neuropathies percentage for each hand | After each cycle (except the 1st one), (each cycle is 7 days)
  Evaluation using the NPSI questionnaire
Cohort 2: Evaluation of the peripheral neuropathies percentage for each hand | At the end of oxaliplatine administration (4 to 6 months after inclusion)
  Evaluation using the NPSI questionnaire
Cohort 2: Evaluation of the peripheral neuropathies percentage for each hand | 12 months after the end of treatment.
  Evaluation using the NPSI questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Thomas BACHELOT, MD, Principal Investigator — Centre Leon Berard
Locations (2):
- France (2):
  - Infirmerie Protestante, Caluire-et-Cuire
  - Centre Léon Bérard, Lyon

REFERENCES:
- [Derived] Hanvic B, Joureau-Chabert A, Ouldbey Y, Toussaint P, Chanel E, Blanc E, Heudel P, Montagnier V, Perol D, Bachelot T. Compression therapy with surgical gloves compared to cold therapy with frozen gloves in preventing paclitaxel-induced peripheral neuropathy: Results from the prospective ELEGANT trial in patients with breast cancer. Eur J Cancer. 2025 Oct 16;229:115791. doi: 10.1016/j.ejca.2025.115791. Epub 2025 Sep 12. PMID 40961808